CLINICAL TRIAL: NCT01793987
Title: The Effect of Coblation on Blood Loss in Endoscopic Sinus Surgery: A Randomized Controlled Trial
Brief Title: Coblation in Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Brian Rotenberg, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BWR001
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Blood Loss
Keywords: blood loss between two groups
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control: shaver (No Intervention)
- Coblation polypectomy (Experimental)
  Interventions: Device: Coblation polypectomy

INTERVENTIONS:
Device: Coblation polypectomy
  Arms: Coblation polypectomy

SUMMARY:
Chronic Rhinosinusitis (CRS) refers to a pathological condition where the sinonasal mucosa is inflamed for greater than 12 weeks(1). It is associated with a constellation of symptoms, including facial pain, anosmia, and nasal congestion. It has been estimated that CRS affects close to 5% of the Canadian population(2). When medical therapy fails, patients are often referred to Otolaryngology- Head and Neck Surgeons for consideration of surgical management. Endoscopic sinus surgery (ESS) is one of the mainstays of therapy for CRS that has failed medical management(3). Traditionally, the microdebrider has been the go-to tool for performing these surgeries, but recently the Coblator (ArthroCare, Austin, Texas) has begun to define its' role in surgery. By using bipolar radiofrequency energy to ablate tissue (with temperatures up to 60˚ C)(4), theoretically the Coblator will result in less bleeding than so-called "cold" surgical techniques (i.e. the microdebrider). In a retrospective study by Eloy et. al, patients with CRS and nasal polyposis had a statistically significant amount of less intraoperative blood loss when the Coblator was used in their surgery, than those patients who underwent surgery with the microdebrider. The investigators plan to further investigate this in a randomized, controlled fashion

ELIGIBILITY:
Inclusion Criteria:

* between 18-70 years old, and
* having a diagnosis of CRS.

Exclusion Criteria:

* previous Endoscopic Sinus Surgery,
* coagulopathies,
* being pregnant, or
* being prescribed anti-coagulants or anti-platelet agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Blood loss | intra-operative

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada